CLINICAL TRIAL: NCT06702189
Title: The Effects of EXOPULSE Mollii Suit on Low Back Pain (EXOBACK)" / EXOPULSE Mollii Suit and Low Back Pain (EXOBACK)
Brief Title: The Effects of EXOPULSE Mollii Suit on Low Back Pain
Acronym: EXOBACK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut De La Colonne Vertebrale Et Des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-A00020-47
Record Dates: First submitted 2024-11-02; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: EXOPULSE Mollii Suit and Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: We designed a randomized, sham-controlled, double-blind trial to demonstrate the improvement of pain, pain-related disability, quality of life, fatigue and mood in adult patients with chronic low back pain following a 2-week intervention of "active" versus "sham" EXOPULSE Mollii suit. A 2-week washout period should be enough to prevent a potential carry-over effect. After this phase (phase 1), a second open-label phase (phase 2) will be proposed for patients to understand the effects of the EXOPULSE Mollii suit employed for 4 weeks (7 sessions per week) on the studied outcomes.
  Summary:
  * Phase 1: randomized sham-controlled crossover study (active versus sham condition)
  * Phase 2: Open-label study (active condition)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Condition (Active Comparator): Active sessions will last 1 hour each. The following parameters will be used for electric stimulation: low frequency (20 Hz), low current intensity (2 mA), with a small pulse width of 25-170 microseconds. These parameters were previously found to be safe in human studies. Based on the clinical exam of each patient, the spastic muscles will be targeted.
  Interventions: Device: EXOPULSE MOLLII SUIT (active)
- Control Condition (Sham Comparator): The control arm will be a sham intervention. The patients will receive a sham stimulation, for which the same EXOPULSE Mollii suit will be used but the suit control unit will be programmed to start stimulating for 1 minute then it will shut off which could enable cutaneous sensations that mimic the active condition, aiming to achieve an effective blinding integrity. There is no risk related to the sham intervention since it consists of applying the same parameters used for the active session (low frequency: 20 Hz; current intensity: 2 mA; pulse width ranging from 25 to 175 µs) but for a shorter duration of time (1 minute).
  Interventions: Device: EXOPULSE MOLLII SUIT (sham)

INTERVENTIONS:
Device: EXOPULSE MOLLII SUIT (active) — Exopulse Mollii suit is a new assistive device that has been developed by Exoneural Network (initially Inerventions AB), a Swedish med-tech company.
  Exopulse Mollii suit is a full-body garment with integrated 58 electrodes that can transcutaneously stimulate several groups of muscles. The device is CE labelled and is intended to use for reducing spasticity and improving blood circulation. The outfit is very easy to put on, it can be used for one hour every day and the analgesic effects last 24 hours or more. EXOPULSE Mollii suit consists of transcutaneous stimulation of several muscles by means of a feeble electric current (i.e., low frequency ~20 Hz, low-intensity 2mA), aiming to reduce pain.
  This treatment method theoretical background primarily refers to the theory of gate control. Based on this theory, the stimulation of large proprioceptive fibers would inhibit the nociceptive information transmitted by small fibers.
  Arms: Experimental Condition
Device: EXOPULSE MOLLII SUIT (sham) — It consists of applying the same parameters used for the active session (low frequency: 20 Hz; current intensity: 2 mA; pulse width ranging from 25 to 175 µs) but for a shorter duration of time (1 minute).
  Arms: Control Condition

SUMMARY:
Low back pain is a common musculoskeletal problem. It is the main cause of activity limitation and work absence and carries a huge medical burden and economic cost. Low back pain is considered "chronic" when it persists for more than 3 months. Chronic low back pain affects daily activities and constitutes a psychological burden, which could lead to anxiety and/or depression. Prevention of low back pain is recognized as a pivotal challenge in high-risk populations to help tackle high healthcare costs related to therapy and rehabilitation. Current pharmacological drugs, namely anti-inflammatory and narcotics medications, have limited efficacy and numerous side effects. In addition, most available treatment options only address single, targeted causes; however, given the complexity of low back pain, a multi-modal interdisciplinary approach is highly needed. Transcutaneous electrical nerve stimulation (TENS) is a safe alternative to current treatments. Many studies have shown its efficacy and benefit in reducing pain. However, it only targets a limited number of muscles. For this reason, transcutaneous stimulation using the EXOPULSE Mollii suit might help reduce pain and related outcomes in this context since it simultaneously targets several muscle groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years, with a definite diagnosis of Low Back Pain for at least 3 months, with absence of any surgical indication.
* Stable pharmacological treatment over the last three months
* Residual back pain post-spinal surgery with no new surgical indication
* Patients should be French speakers, able to understand verbal instructions, and affiliated to the national health insurance NHI.

Exclusion Criteria:

* Patient with VAS < 4
* Presence of any surgical indication (i.e,. isthmic spondylolisthesis, herniated disc, Spinal canal stenosis, Vertebral fracture, Degenerative Spondylolisthesis, scoliosis)
* Failed Back Surgery Syndrome (FBSS)
* Presence of spinal infection
* Presence of obstetrical or gynecological cause of the low back pain (ovarian torsion, ovarian cyst, endometriosis, menses)
* Retroperitoneal tumors - Spinal tumors - Being included in another research protocol during the study period
* Inability to undergo medical monitoring for the study purposes due to geographical or social reasons
* Having a cardiac stimulator, a ventriculoperitoneal shunt, an intrathecal baclofen pump, or other contraindications to using EXOPULSE Mollii suit
* Being pregnant
* Having a change in their pharmacological therapy in the last three months.
* Suffering from other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain)
* Having a body mass index above 35 Kg/m2
* In case of the introduction of a medical device other than EXOPULSE Mollii suit during the study period
* Patients under juridical protection (" mesure de protection judiciaire : tutelle, curatelle, sauvegarde de justice ")
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain-related disability reduction will be assessed using the QBPDS (Quebec Back Pain Disability Scale) before and after active and sham stimulation | This will be assessed through study completion, an average of 3 months at Visit 1(Day 0) , Visit 2 (Day 15), Visit 3 (Day 30), Visit 4 (Day45), Visit 5 (Day 60) and Visit 6 (Day 90)
  The QBPDS (Quebec Back Pain Disability Scale) is a 20-item scale that is widely used in back pain research. Items evaluate the ability to perform the mentioned activity and are rated using 5 possibilities ranging from "not difficult at all" to "unable to do". Lower scores reflect lower disability. The French version has good psychometric properties (internal consistency, content validity, and acceptability).

SECONDARY OUTCOMES:
Assessment of pain-related disability reduction using the ODQ (Owestry Disability scale) | This will be assessed through study completion, an average of 3 months (at Visits 1, 2, 3, 4, 5 and 6)
  The ODQ (Owestry Disability scale) consists of 10 items questionnaire (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, driving/riding a car, changing degree of pain) rated using 6 possibilities as well as a visual item assessing pain quality from absence to extreme. ). Lower scores reflect lower disability.
Analgesic effects based on the VAS (Visual Analogue Scale) | This will be assessed through study completion, an average of 3 months (at Visits 1, 2, 3, 4, 5 and 6)
  The visual analogue scale of pain (VASpain) consists of rating the symptom on a 10 cm horizontal line going from "no pain" to "worst pain imaginable" .
Analgesic effects based on the Brief Pain Inventory (BPI) | This will be assessed through study completion, an average of 3 months (at Visits 1, 2, 3, 4, 5 and 6)
  The validated French version of the Brief Pain Inventory (BPI) will be used to assess pain severity (4 items) and pain interference (7 items). BPI items are rated on a 10-point scale running from 0 (no pain/does not interfere) to 10 (pain as bad as you can feel/interferes completely). A total pain severity score can be found by averaging these items. Higher scores indicate greater severity and more interference.
Analgesic effects based on the Pain Catastrophizing Scale (PCS) | This will be assessed through study completion, an average of 3 months (at Visits 1, 2, 3, 4, 5 and 6)
  The Pain Catastrophizing Scale (PCS) is a valid and reliable scale that includes 13 items assessing the presence and severity of feelings or thoughts that emerge when experiencing pain. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time). Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Assessment of anti-fatigue effects according to VAS (visual analogue scale) | This will be assessed through study completion, an average of 3 months (at Visits 1, 2, 3, 4, 5 and 6)
  The visual analogue fatigue scale (EVA fatigue) is a 10 mm straight hozontal line, with one end corresponding to no fatigue and the other to extreme fatigue.
Mood symptoms will be evaluated using the Hospital Anxiety and Depression Scale (HADS) | This will be assessed through study completion, an average of 3 months (at Visits 1, 2, 3, 4, 5 and 6)
  It is a 14-item generic scale with good psychometric properties. It consists of seven items assessing anxiety and seven others assessing depression. Scores can range from 0 to 21 on each subscale, with higher scores indicating worse symptomatology .
Improvement of the quality of life using the Short Form 36 Health Survey (SF-36) | This will be assessed through study completion, an average of 3 months (at Visits 1, 2, 3, 4, 5 and 6)
  It is a generic survey that contains 36 items that assess the quality of life and yield eight dimensions: physical functioning, physical role, emotional role, bodily pain, general health, vitality, social functioning, and mental health. The score of each dimension ranges from 0 to 100, with higher scales implying better health status. The French version has excellent convergent and discriminant validity (100% and 97.9%, respectively) and good internal consistency.
Evaluation of overall improvement using the CGI (Clinical Global Impression) | This will be assessed at Visit2 (Day 15) , Visit4 (Day 45) and Visit6 (Day 90) since CGI is designed to be applied after interventions
  It consists of 7-point scale ranging from "very much improved since the initiation of treatment" to "very much worse since the initiation of treatment" (from 1 to 7)
Evaluation of patient's blinding to the type of stimulation in the crossover trial | This will only be assessed at Visit2 (Day 15) and Visit4 (Day 45) of Phase 1.
  This blind evaluation will be done in phase 1 using a dedicated questionnaire (only for each condition since all patients will receive the same active treatment in the open-label phase 2).

CONTACTS AND LOCATIONS:
Overall Officials: Samar S Ayache, MD, PhD, HDR, Principal Investigator — Hopital Henri Mondor, Assistance Publique - Hôpitaux de Paris, Créteil, France
Locations (1):
- Clinical Neurophysiology department, Henri Mondor Hospital, Créteil, France, Créteil, VAL DE MARNE, France